CLINICAL TRIAL: NCT00148642
Title: Multi-center Clinical Trial of the Bard Silver-coated Endotracheal Tube to Reduce Ventilator Associated Pneumonia (VAP)
Brief Title: Silver-Coated Endotracheal Tube to Reduce Ventilator Associated Pneumonia (VAP)
Acronym: NASCENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Joan Dulin, CR Bard, Inc
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 5003A
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Respiratory Failure
Keywords: ventilator-associated pneumonia; nosocomial pneumonia
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): silver salts coated endotracheal tube
  Interventions: Device: silver salts coated endotracheal tube
- 2 (Placebo Comparator): uncoated endotracheal tube
  Interventions: Device: uncoated endotracheal tube

INTERVENTIONS:
Device: silver salts coated endotracheal tube — intubation with silver coated tube
  Other Names: Agento
  Arms: 1
Device: uncoated endotracheal tube — intubation
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the use of a silver-coated endotracheal tube (ETT) can reduce the incidence and/or delay the time of onset of VAP when compared to a non silver-coated ETT in patients who have been mechanically ventilated for >= 24 hours.

DETAILED DESCRIPTION:
Nosocomial pneumonia is the leading cause of death from hospital-acquired infections.Ventilator associated pneumonia (VAP) develops in a significant percentage of patients who have been ventilated for at least 48 hours, and is associated with high morbidity, mortality,and financial costs. Silver is a well-characterized antimicrobial agent, and is the active agent in multiple medical products used to reduce or control infection. Bard has developed a proprietary antimicrobial ETT, manufactured with a hydrophilic coating containing a fine dispersion of silver salts.

This study compare the incidence and time to onset of VAP in patients intubated for >=24 hours with a proprietary silver-coated ETT versus those intubated for >= 24 hours with a standard non-coated ETT.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* expected to be intubated for at least 24 hours
* able to sign Informed Consent

Exclusion Criteria:

* symptoms of bronchiectasis
* severe hemoptysis
* history of cystic fibrosis
* intubated > 12 hours within previous 30 days
* pregnancy
* participating in a competing trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2003 (Actual)
Dates: Start 2002-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The incidence of microbiologically-confirmed VAP (mVAP), as determined by quantitative culture of bronchoalveolar lavage fluid, in subjects intubated for >=24 hours. | 30 days

SECONDARY OUTCOMES:
time to onset of mVAP in subjects intubated for >=24 hours | 30 days
incidence of clinical VAP in subjects intubed for >=24 hours | 30 days
duration of intubation | unlimited
mortality | unlimited
antibiotic usage | unlimited
length of stay | unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Marin H Kollef, MD, Principal Investigator — Barnes Jewish Hospital, St. Louis, MO
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - West Suburban Hospital, Oak Park, Illinois
  - Mayo Clinic & Foundation, Rochester, Minnesota
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Audie Murphy VA Medical Center & University Hospital, San Antonio, Texas

REFERENCES:
- [Background] Baughman RP, Spencer RE, Kleykamp BO, Rashkin MC, Douthit MM. Ventilator associated pneumonia: quality of nonbronchoscopic bronchoalveolar lavage sample affects diagnostic yield. Eur Respir J. 2000 Dec;16(6):1152-7. doi: 10.1034/j.1399-3003.2000.16f23.x. PMID 11292122
- [Derived] Restrepo MI, Anzueto A, Arroliga AC, Afessa B, Atkinson MJ, Ho NJ, Schinner R, Bracken RL, Kollef MH. Economic burden of ventilator-associated pneumonia based on total resource utilization. Infect Control Hosp Epidemiol. 2010 May;31(5):509-15. doi: 10.1086/651669. PMID 20302428
- [Derived] Kollef MH, Afessa B, Anzueto A, Veremakis C, Kerr KM, Margolis BD, Craven DE, Roberts PR, Arroliga AC, Hubmayr RD, Restrepo MI, Auger WR, Schinner R; NASCENT Investigation Group. Silver-coated endotracheal tubes and incidence of ventilator-associated pneumonia: the NASCENT randomized trial. JAMA. 2008 Aug 20;300(7):805-13. doi: 10.1001/jama.300.7.805. PMID 18714060